CLINICAL TRIAL: NCT02619266
Title: The Traditional Chinese Medicine Department of Xin Qiao Hospital
Brief Title: The Safety and Effect Study of Acupuncture for Anorexia in Patients With Gastrointestinal Tract and Lung Cancers
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chaoting Zhao, Vice Director, Clinical Reseach, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014YLC32; 2015CB554504 (Other Grant/Funding Number: National Program on Key Basic Research Project (973 Program))
Record Dates: First submitted 2015-11-23; First posted 2015-12-02 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Anorexia; Cancer Cachexia
Keywords: Cancer Anorexia Cachexia Syndrome; Acupuncture; Megestrol acetate; Poor Appetite; Anorexia; Randomized Controlled Trial
MeSH Terms: conditions — Anorexia | interventions — Acupuncture Therapy; Megestrol Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acupuncture+Placebo (Experimental): Acupuncture once daily for 7 days and Placebo tablet by mouth, twice a day for 7 days.
  Interventions: Other: Acupuncture; Drug: Placebo(Megestrol Acetate)
- Megestrol Acetate+Sham acupuncture (Active Comparator): Megestrol Acetate tablet 160mg by mouth, twice a day for 7 days and Sham Acupuncture once a day for 7 days .
  Interventions: Other: Sham Acupuncture; Drug: Megestrol Acetate
- Placebo+Sham acupuncture (Placebo Comparator): Placebo tablet by mouth, twice a day for 7 days and Sham Acupuncture once a day for 7 days .
  Interventions: Other: Sham Acupuncture; Drug: Placebo(Megestrol Acetate)

INTERVENTIONS:
Other: Acupuncture — Acupuncture is the practice of inserting thin needles into specific points to improve health and well-being.
  Other Names: Real acupuncture; True acupuncture
  Arms: Acupuncture+Placebo
Other: Sham Acupuncture — Sham acupuncture is used as a control in scientific studies that test the efficacy of acupuncture in the treatment of various illness or disorders.
  Arms: Megestrol Acetate+Sham acupuncture; Placebo+Sham acupuncture
Drug: Megestrol Acetate — Megestrol Acetate 160mg tablet
  Other Names: Positive Drug
  Arms: Megestrol Acetate+Sham acupuncture
Drug: Placebo(Megestrol Acetate) — Starch pill manufactured to mimic Megestrol Acetate 160mg tablet
  Other Names: Placebo Pill
  Arms: Acupuncture+Placebo; Placebo+Sham acupuncture

SUMMARY:
This trail will be carried out to evaluated the effect and safety of acupuncture for the anorexia in patients with gastrointestinal tract and lung cancers.

DETAILED DESCRIPTION:
Acupuncture used for anorexia related to cancer, but there were lack of powerful evidence. The 160 eligibilities will be randomly divided into 3 groups(Acupuncture and Placebo group, Megestrol acetate and Sham Acupuncture group, Placebo and Sham Acupuncture group).The effect will be investigated baseline, the 2,5,8 and 15days. The safety issue will be recorded every section during the acupuncture.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed gastrointestinal tand lung cancers;
2. Age ≥18 years;
3. Appetite score≤ 6 (0= worst appetite), and the symptom lasted 2 weeks at lest at screening;
4. Had a history of weight loss ≥5% within 6 moths;
5. Maintained oral intake;
6. Signed the informed consent.

Exclusion Criteria:

1. Patients with dementia, delirium, intestinal obstruction, pregnancy or lactation;
2. Had uncontrolled symptoms that could impact appetite or caloric intake such as nausea, pain, or depression(The score of the symptoms≤ 3, 0= worst) ;
3. Patients with untreated vitamin B12 deficiency or endocrine abnormalities(thyroid dysfunction and hypoadrenalism);
4. Patients on melatonin supplements or medications with potential appetite-stimulating activity(Chinese herb,thalidomide)
5. Less than one week before the screening or there will be a surgery ,radiotherapy and chemotherapy the acupuncture;
6. Lifetime expected less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Appetite Visual Analog Scale | Baseline, the days 8 and 15.
  The assessment will be done thirty minutes before meals. The participators should record the score of their appetite (0 to 100 mm) the higher scores reflect better symptom control.

SECONDARY OUTCOMES:
Council of Nutrition appetite questionnaire (CNAQ) | Baseline, the days 8 and 15.
  Ask the subjects to complete the questionnaire by circling the correct answers and then tally the results based upon the following numerical scale: a =1, b = 2, c = 3, d = 4, e = 5. The sum of the scores for the individual items constitutes the CNAQ score. CNAQ score ≤28 indicates significant risk of at least 5% weight loss within six months.
Caloric intake | Baseline, the days 8 and 15.
  The caloric intake will be assessed by the dietician.
Functional Assessment of Anorexia/Cachexia Therapy | Baseline, the days 8 and 15.
  Functional Assessment of Anorexia/Cachexia Therapy was designed to measure general aspects of quality of life (QOL) as well as specific anorexia/cachexia-related concerns.
Nutritional status | Baseline, the days 8 and 15.
  weight was determined in kilograms. Triceps skinfold (mm), arm circumference(cm), and calf circumference (cm) were determined

OTHER OUTCOMES:
Edmonton Symptom Assessment Scale | Baseline, the days 8 and 15.
  Edmonton Symptom Assessment Scale is a nine-item patient-rated symptom visual analogue scale developed for use in assessing the symptoms of patients receiving palliative care.
The Questionnaire of Acupuncture-related Events(QAE) | Baseline and the days 7
  The side effects and their detail will be record during and after the acupuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Tang, PhD, Study Chair — Chengdu University of Traditional Chinese Medicine; Chaoting Zhao, MD, Study Director — Xinqiao Hospital; Haiou Luo, PhD, Principal Investigator — Xinqiao Hospital
Locations (4):
- China (4):
  - Chongqing TCM Hospital, Jiangbei, Chongqing Municipality
  - XinQiao Hosiptal, Shapingba, Chongqing Municipality
  - Donghua Hosiptal, Shapingba, Chongqing Municipality
  - Daping Hospital, Yuzhong, Chongqing Municipality

REFERENCES:
- [Background] Del Fabbro E, Dev R, Hui D, Palmer L, Bruera E. Effects of melatonin on appetite and other symptoms in patients with advanced cancer and cachexia: a double-blind placebo-controlled trial. J Clin Oncol. 2013 Apr 1;31(10):1271-6. doi: 10.1200/JCO.2012.43.6766. Epub 2013 Feb 25. PMID 23439759
- [Background] Bruera E, Strasser F, Palmer JL, Willey J, Calder K, Amyotte G, Baracos V. Effect of fish oil on appetite and other symptoms in patients with advanced cancer and anorexia/cachexia: a double-blind, placebo-controlled study. J Clin Oncol. 2003 Jan 1;21(1):129-34. doi: 10.1200/JCO.2003.01.101. PMID 12506181
- [Background] Bruera E, Macmillan K, Kuehn N, Hanson J, MacDonald RN. A controlled trial of megestrol acetate on appetite, caloric intake, nutritional status, and other symptoms in patients with advanced cancer. Cancer. 1990 Sep 15;66(6):1279-82. doi: 10.1002/1097-0142(19900915)66:63.0.co;2-r. PMID 2205358
- See also: Acupuncture for Unintentional Weight Loss and Anorexia With GI Cancer — http://www.clinicaltrials.gov/ct2/show/NCT02148159